CLINICAL TRIAL: NCT02247765
Title: Controlled Acute Hypoxia Study Comparing Pulse Oximetry to Arterial Blood Samples During Motion in Healthy, Well Perfused Subjects With the USB Pulse Oximetry Monitor Interface Cable
Brief Title: Controlled Acute Hypoxia Study Comparing Pulse Oximetry to Arterial Blood Samples During Motion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: COVMOPR0445
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Healthy; Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arterial Line (Experimental): CO-Oximetry value obtained as a comparator. Obtained during motion conditions.
  Interventions: Device: Arterial line
- Motion (Experimental): The subject has to perform motions during the procedure. This is to verify that device is able to read through motion.
  Interventions: Device: Motion

INTERVENTIONS:
Device: Arterial line — Arterial line is inserted to draw a CO-Oximeter value as it is the gold standard and as advised in ISO 80601
  Other Names: CO-Oximeter SaO2 value
  Arms: Arterial Line
Device: Motion — The subject is asked to move their hand by either rubbing or tapping their fingers at a specified frequency and amplitude during portions of the hypoxic procedure.
  Arms: Motion

SUMMARY:
To validate the proposed claims for pulse rate and saturation accuracy in a diverse subject population during motion over a specified saturation range.

DETAILED DESCRIPTION:
Use an investigational oximetry system to evaluate the triggering of the "sensor off" status with marketed, off-the-shelf sensors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race
* 18-50 years old, inclusive
* Females: negative urine pregnancy test on the day of study participation (prior to exposure to hypoxia)
* Completed within the last year: physical exam by a licensed physician, physician assistant (PA), or advanced practice nurse; including a 12 lead ECG, a medical history, and blood test (complete blood count and sickle cell trait/disease screening)
* Meets specific demographic requirements for the monitoring device under study
* Willing and able to provide written informed consent
* Able to participate for the duration of the evaluation

Exclusion Criteria:

* A room-air baseline % modulation < 1.5% on all four fingers on the test hand
* Under 18 years or over 50 years of age
* Pregnant and/or lactating women
* Hypertension: on three consecutive readings, systolic pressure greater than 145 mm Hg or diastolic pressure greater than 90 mm Hg
* Ventricular premature complexes (VPC's) that are symptomatic or occur at a rate of more than four per minute
* History of seizures (except childhood febrile seizures) or epilepsy
* History of unexplained syncope
* Daily or more frequent use of anxiolytic drugs (benzodiazepines) for treatment of anxiety disorder
* Recent history of frequent migraine headaches: average of two or more per month over the last year
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* History of acute altitude sickness at or below moderate elevation (up to 5,000-10,000 feet) defined as three or more of the following symptoms: moderate to severe headache, general malaise, dizziness/lightheadedness, nausea/vomiting, fatigue/weakness, shortness of breath, nosebleed, persistent rapid pulse, or peripheral edema
* History of significant respiratory disease such as severe asthma or emphysema or sleep apnea
* Sickle cell disease or trait
* Clinically significant abnormal finding on medical history, physical examination, clinical laboratory test or ECG. Clinical significance will be assessed by the principal investigator or study physician as designated.
* History of stroke, transient ischemic attack or carotid artery disease
* History of myocardial ischemia, angina, myocardial infarction, congestive heart failure or cardiomyopathy
* History of chronic renal impairment
* Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
* Unwillingness or inability to remove colored nail polish or artificial nails from test digit(s)
* Unwillingness or inability to give informed consent
* Prior or known allergies to: lidocaine (or similar pharmacological agents, e.g., Novocain) or heparin
* Recent arterial cannulation (i.e., less than 30 days prior to study date)
* Six or more arterial cannulations of each (right & left) radial artery
* History of clinically significant complications from previous arterial cannulation
* Current use of blood thinners: prescription or daily aspirin use
* History of bleeding disorders or personal history of prolonged bleeding from injury.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Heyer, MD, Principal Investigator — Medtronic - MITG
Locations (2):
- United States (2):
  - Boulder Clinical Laboratory, Boulder, Colorado
  - Covidien RMS, Boulder, Colorado

RESULTS

PARTICIPANT FLOW:
Groups:
- USB Pulse Oximetry Monitor Interface Cable: Additional interventions include the following: Radial Arterial Line placement involves introduction of a standard arterial catheter or angiocath into the radial artery. Since the arterial catheter is placed into the artery using a needle, there will be mild to moderate discomfort. The total amount of blood drawn during the procedure is less than 100cc.
  Additionally, subjects are asked to perform motions with their hand. Standard motions include tapping and rubbing at aperiodic intervals with amplitudes of 1-2 cm and 1-4 Hz with a random variation in frequency. The subject is instructed to tap (or rub) with finger tips to maintain consistency of area of effect on the pressure pad and to prevent resting hand on pressure pad between motions so that only qualified taps are recorded by the pressure pad system. Each plateau will have both an interval of tapping and rubbing.
Period: Overall Study
Arm/Group | USB Pulse Oximetry Monitor Interface Cable
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | no Treatment
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.67 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: SpO2 Accuracy During Motion Conditions - MaxA Sensor
Description: For each range specified, SpO2 accuracy of the pulse oximeter equipment is stated in terms of the Accuracy Root-Mean-Square (ARMS) difference between measured values (SpO2) and reference blood values (SaO2). The MaxA sensors has a different bandage from the MaxN sensor, and therefore a different form and fit.
Time Frame: up to 6 months
Measure: Number; unit: Accuracy Root Mean Square
Arm/Group | no Treatment
Number analyzed (Participants) | 18
Accuracy Root Mean Square | 1.78

2. Primary Outcome: SpO2 Accuracy During Motion Conditions - MaxN Sensor
Description: For each range specified, SpO2 accuracy of the pulse oximeter equipment is stated in terms of the Accuracy Root-Mean-Square (ARMS) difference between measured values (SpO2) and reference blood values (SaO2). The MaxN sensor has a different bandage from the MaxA sensor, and therefore a different form and fit.
Time Frame: up to 6 months
Measure: Number; unit: Accuracy Root Mean Square
Arm/Group | no Treatment
Number analyzed (Participants) | 18
Accuracy Root Mean Square | 1.93

ADVERSE EVENTS:
Arm/Group | no Treatment
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | no Treatment (N=18)
mild IV infiltration (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No